CLINICAL TRIAL: NCT05295459
Title: ENLIGHTEN 2: A Phase III, Randomized, Blinded, Controlled, Parallel-Group Trial to Evaluate the Efficacy and Safety of LYR-210 for the Treatment of Chronic Rhinosinusitis in Adults
Brief Title: Efficacy and Safety of LYR-210 for the Treatment of Chronic Rhinosinusitis in Adults (ENLIGHTEN 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lyra Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYR-210-2021-005
Record Dates: First submitted 2022-03-08; First posted 2022-03-25 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Chronic Sinusitis; Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LYR-210 (Experimental): Single administration of LYR-210 drug matrix (7500 μg)
  Interventions: Drug: LYR-210; Other: Background therapy
- Sham procedure control (Sham Comparator): Single mock administration procedure
  Interventions: Drug: Sham procedure control; Other: Background therapy

INTERVENTIONS:
Drug: LYR-210 — LYR-210 drug matrix (mometasone furoate)
  Arms: LYR-210
Drug: Sham procedure control — Sham procedure control
  Arms: Sham procedure control
Other: Background therapy — Daily Saline Irrigation

SUMMARY:
Multicenter, phase III, randomized, blinded, controlled, parallel group.

DETAILED DESCRIPTION:
This is a 24-week, multicenter, phase III, randomized, blinded, controlled, parallel group with a 24-week treatment period to evaluate the efficacy and safety of LYR-210 compared with sham control for treatment in adults with CRS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Diagnosed as having CRS
* Bilateral ethmoid disease confirmed on CT
* Mean 3 cardinal symptom (3CS) score
* Undergone at least 2 trials of medical treatments in the past
* Has been informed of the nature of the study and provided written informed consent
* Agrees to comply with all study requirements
* If currently on a waiting list for sinonasal surgery, willing to be removed from the waiting list or have preplanned surgery date cancelled for the duration of the study. [Note: this does not preclude a participant from receiving or being recommended for sinonasal surgery as rescue treatment during the study].

Exclusion Criteria:

* Inability to tolerate topical anesthesia
* Previous nasal surgery
* Presence of nasal polyp grade 2 or higher
* Seasonal allergic rhinitis
* Perennial rhinitis with symptoms that are well controlled by regular use of intranasal corticosteroids
* Severe asthma
* History or clinical evidence or suspicion of invasive fungal sinusitis, allergic fungal rhinosinusitis, atrophic rhinitis, or odontogenic sinusitis
* Obstruction preventing proper placement and retention of LYR-210 as seen on endoscopy
* Anatomic variation that, in the opinion of the investigator, would adversely impact placement of LYR-210 as seen on CT
* Known history of hypersensitivity or intolerance to corticosteroids
* Known history of hypothalamic pituitary adrenal axial dysfunction
* Previous pituitary or adrenal surgery
* Dental procedure/implant on maxillary dentition within 4 weeks of the Screening visit.
* Past or present acute or chronic intracranial or orbital complications of CRS
* History or diagnosis (in either eye) of glaucoma or ocular hypertension
* Past or present functional vision in only 1 eye
* Past, present, or planned organ transplant or chemotherapy with immunosuppression
* Currently positive for COVID-19 or residual sinonasal symptoms from a previous COVID-19 infection
* Pregnant or breast feeding. Females of child-bearing potential must test negative for pregnancy at the time of screening
* Evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments
* Currently participating in an investigational drug or device study
* Determined by the investigator as not suitable to be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline (CFBL) in the 7-day average composite score of 3 cardinal symptoms (3CS) of nasal blockage/obstruction/congestion, anterior/posterior nasal discharge, and facial pain/pressure at Week 24 in participants without nasal polyps. | Week 24
  The 3CS are nasal blockage/obstruction/congestion, anterior/posterior nasal discharge, and facial pain/pressure. Each symptom is rated on a 4-point (0-3) scale where 0=absent symptoms and 3=severe symptoms. The composite score of 3CS is the sum of the three cardinal symptom scores.

SECONDARY OUTCOMES:
CFBL in the 7-day average composite score of 3CS at Week 24. | Week 24
  The 3CS are nasal blockage/obstruction/congestion, anterior/posterior nasal discharge, and facial pain/pressure. Each symptom is rated on a 4-point (0-3) scale where 0=absent symptoms and 3=severe symptoms. The composite score of 3CS is the sum of the three cardinal symptom scores.
CFBL in the 22-item Sino-Nasal Outcome Test (SNOT-22) total score at Week 24. | Week 24
  The SNOT-22 questionnaire is a 22-item disease-specific quality of life instrument. Each symptom is scored on a 6-point scale where 0 = no problem and 5 = problem as bad as it can be. The total SNOT-22 score is the sum of the 22 items and can range from 0 to 110 with higher scores indicating worse symptoms.
CFBL in the percent opacification of the bilateral anterior and posterior ethmoids at Week 20, as determined by 3-D volumetric CT analysis. | Week 20
  Change from baseline in the 3-D volumetric CT score at Week 20.
Rescue treatment requirement through Week 24. | Week 24
  Number and percent of participants requiring rescue treatment through Week 24, this data will be conducted from pooled data from Enlighten 2 and the Enlighten I study.

CONTACTS AND LOCATIONS:
Locations (57):
- United States (31):
  - Novak Clinical Trials, Tucson, Arizona
  - Keck School of Medicine at USC Medical Center, Arcadia, California
  - Sensa Health Clinical Research, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California - Irvine Medical Center, Orange, California
  - Sacramento Ear Nose and Throat Surgical and Medical Group, Inc, Roseville, California
  - University of California - Davis, Sacramento, California
  - Regional Head & Neck Consulting - SENTA Clinic, San Diego, California
  - Breathe Clear Institute, Torrance, California
  - Colorado ENT and Allergy, Colorado Springs, Colorado
  - Ear, Nose and Throat Associates of South Florida, P.A., Boynton Beach, Florida
  - ENT and Allergy Associates of Florida - Brandon, Brandon, Florida
  - ENT and Allergy Associates of Florida - Plantation - Dr. Johnson, Plantation, Florida
  - ENT and Allergy Associates of Florida - Plantation - Dr. Wright, Plantation, Florida
  - ENT and Allergy Associates of Florida, Port Saint Lucie, Florida
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center (KUMC), Fairway, Kansas
  - Tandem Clinical Research, Marrero, Louisiana
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - University of Missouri-Columbia, Columbia, Missouri
  - St Louis University, St Louis, Missouri
  - ENT and Allergy Associates, LLP - Fifth Avenue New York, New York, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - ENT and Allergy Associates - White Plains, White Plains, New York
  - Carolina Ear, Nose, & Throat Clinic/CENTRI, Inc., Orangeburg, South Carolina
  - Houston Methodist Hospital, Houston, Texas
  - ENT Associates of Texas, McKinney, Texas
  - Lyra Investigational Site, Ogden, Utah
  - Lyra Investigational Site, Richmond, Virginia
- Belgium (2):
  - University Hospital Gent, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
- Bulgaria (4):
  - University Multiprofile Hospital for Active Treatment, Burgas
  - UMHAT Kaspela Ltd, Plovdiv
  - Military Medical Academy Multiprofile Hospital, Sofia
  - Diagnostic and Consulting Center Mladost - Varna, Varna
- Germany (5):
  - HNO Praxis Dr. Andrea Kienle-Gogolok, Baden
  - HNO Zentrum am Kudamm, Berlin
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - HNO Landsberg, Landsberg
  - Universitaetsklinikum Tuebingen, Tübingen
- Hungary (8):
  - Semmelweis Egyetem - Nyaksebeszeti Klinika, Budapest
  - Budapesti Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Szent Imre Korhaz, Budapest
  - Eszak-Pesti Centrumkorhaz - Honvedkorhaz, Budapest
  - Budapesti Uzsoki Utcai Korhaz, Budapest
  - Lyra Investigational Site, Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz, Tatabánya
- Poland (7):
  - Sleepmedica, Bialystok
  - "Farma-Med." Kujawskie Centrum Medyczne Sp. z o.o., Inowrocław
  - Promed P.Lach R.Glowacki Spolka Jawna, Krakow
  - Velocity Lublin, Lublin
  - Mazowiecki Szpital Brodnowski Sp. z o.o. - Zespol Oddzialow Otolaryngologii, Warsaw
  - Lyra Investigational Site, Warsaw
  - Panstwowy Instytut Medyczny MSWiA - Klinika Otolaryngologii, Wroclaw